CLINICAL TRIAL: NCT04279262
Title: Community First Responders' Role in the Current and Future Rural Health and Care Workforce
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Other Study IDs: 20002
Record Dates: First submitted 2020-01-23; First posted 2020-02-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2022-05

CONDITIONS: Emergency Medical Services
Keywords: Community first responder; Rural health; Ambulance service

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anonymised records from 6 ambulance services: The total available sample for analysis for this cohort is estimated to be at least 50,000 incidents across 6 ambulance trusts. The investigators will describe the epidemiology of CFR provision to rural health areas using an anonymised dataset.
  Interventions: Other: attendance by community first responders for medical emergencies
- Interviews with patients (and/or relatives): The investigators will interview about 15-20 patients (and/or relatives) who have been attended by CFRs.
  Interventions: Other: attendance by community first responders for medical emergencies
- Interviews with CFRs: The investigators will interview about 15-20 CFRs/ CFR scheme leaders.
- Interviews with Ambulance staff: The investigators will interview about 15-20 ambulance staff who have experience of working with CFRs.
- Interviews with GPs and commisioners: The investigators will interview about 10-15 GPs and ambulance service commissioners.

INTERVENTIONS:
Other: attendance by community first responders for medical emergencies — The investigators will purposively sample patients, relatives, and ambulance staff identified from records of patients who have been attended by a CFR in a rural location in the previous six months. Where possible the investigators will interview patients, relatives, CFRs and ambulance staff attending the same event. GPs will be purposively sampled from rural areas of the ambulance services involved. Investigators will recruit a maximum variation sample of patients (according to age, sex, condition, and ethnicity), ambulance staff (sex, experience, ethnicity and role), CFR (sex, ethnicity, length of experience, skill level) and CFR scheme leads (independent charity and ambulance trust overseen schemes).
  Groups: Anonymised records from 6 ambulance services; Interviews with patients (and/or relatives)

SUMMARY:
Community First Responders (CFRs) are trained members of the public, lay people or off-duty healthcare staff who volunteer to provide first aid. CFRs help ambulance services to provide care for people having health emergencies, from falls to road accidents to heart attacks, at home or in public places. CFRs are particularly important in rural areas where it is more difficult to provide or access emergency care, and where they are an important part of the care workforce. CFRs are broadly perceived to be positive, however evidence is needed about how they contribute to rural health services, which patients/conditions they attend, what care they provide, how effective they are and at what cost, how they are perceived by patients and other health workers, and how they could be developed to improve care for rural communities.

The investigators aim to develop recommendations for rural CFRs, by exploring their contribution to rural care, evaluating their value for money, understanding experiences and views of patients, CFRs and other healthcare staff, and exploring the potential for CFRs to provide new services.

DETAILED DESCRIPTION:
The project will involve the following steps:

1. Analyse records from six ambulance services to see: how many people CFRs attended; the proportion of ambulance calls attended; age, sex and conditions of people attended; how quickly CFRs attended and what happened to the patient(s) when the ambulance arrived.
2. Evaluate benefits and costs of CFRs attending rural emergencies.
3. Interview patients/relatives, ambulance staff, GPs, funders, CFRs and CFR leads to obtain views on rural CFR current and potential future roles. Interviews will also explore with CFRs and CFR leads, challenges and solutions to recruiting, training, retaining rural CFRs and ensuring safe, high quality care.
4. Combine this knowledge (gained in steps1-3 above) to develop recommendations for change; who will be involved and how services should change to solve the most pressing problems for the rural communities served.
5. Present recommendations to a workshop of experts and public to agree priorities for future development.

ELIGIBILITY:
Inclusion Criteria:

* Adults capable of giving informed consent. The investigators will recruit a maximum variation sample of patients (according to age, sex, condition, and ethnicity), ambulance staff (sex, experience, ethnicity and role), CFR (sex, ethnicity, length of experience, skill level) and CFR scheme leads (independent charity and ambulance trust overseen schemes).

Exclusion Criteria:

* The investigators will exclude children and adults who are unable to give informed consent from this study.

London Ambulance Service NHS Trust is not included as it is mainly urban; East of England Ambulance Service and North East Ambulance Service are not included because of lack of electronic data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the interview studies the investigators will purposively sample patients, relatives, and ambulance staff identified from records of patients who have been attended by a CFR in a rural location in the previous six months. Where possible the investigators will interview patients, relatives, CFRs and ambulance staff attending the same event. GPs will be purposively sampled from rural areas of the ambulance services involved. The investigators will recruit a maximum variation sample of patients (according to age, sex, condition, and ethnicity), ambulance staff (sex, experience, ethnicity and role), CFR (sex, ethnicity, length of experience, skill level) and CFR scheme leads (independent charity and ambulance trust overseen schemes).
Sampling Method: Non-Probability Sample
Enrollment: 83995 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Number of ambulance calls that CFRs attend in one year | we will evaluate all emergency attendances during one year
  We will establish how many people CFRs attended and work out the proportion of ambulance calls attended.
The type of cases treated by CFRs | we will evaluate all emergency attendances during one year
  characteristics of people (age, sex, condition) attended
How quickly cases are dealt with | we will evaluate all emergency attendances during one year
  how quickly they attend
Treatments given and transfer to hospital | we will evaluate all emergency attendances during one year
  we will evaluate the treatments provided and the number of cases transferred to hospital
Locations | we will evaluate all emergency attendances during one year
  We will describe rurality and location (eg. at home or elsewhere) where CFRs give treatment.

SECONDARY OUTCOMES:
Perceptions of CFR schemes | participants will have been involved in a CFR attendance in the previous 6 months
  We will interview different stakeholders (patients, CFRs, GPs, ambulance staff, CFR leads)

CONTACTS AND LOCATIONS:
Overall Officials: Niro Siriwardena, Principal Investigator — University of Lincoln, UK
Locations (1):
- Community and Health Research Unit, University of Lincoln, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siriwardena AN, Patel G, Botan V, Smith MD, Phung VH, Pattinson J, Trueman I, Ridyard C, Hosseini MP, Asghar Z, Orner R, Brewster A, Mountain P, Rowan E, Spaight R. Community First Responders' role in the current and future rural health and care workforce: a mixed-methods study. Health Soc Care Deliv Res. 2024 Jul;12(18):1-101. doi: 10.3310/JYRT8674. PMID 39054745

DOCUMENTS (1):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT04279262/Prot_000.pdf